CLINICAL TRIAL: NCT06386055
Title: Air Pollution and Physical Activity: A Randomized Controlled Trial
Brief Title: Air Pollution and Physical Activity Study
Acronym: PARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Lina Mu, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00007545
Record Dates: First submitted 2024-04-24; First posted 2024-04-26 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Physical Inactivity; Pollution; Exposure
MeSH Terms: conditions — Sedentary Behavior | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention group 1 (Experimental): This is the physical intervention group 1(n=8).
  Interventions: Behavioral: Active exercise
- Intervention group 2 (Experimental): This is the physical intervention group 2(n=8).
  Interventions: Behavioral: Active exercise
- Control group (No Intervention): This is the control group (n=8).

INTERVENTIONS:
Behavioral: Active exercise — The intervention group will be provided with training courses for 3 months.
  Arms: Intervention group 1; Intervention group 2

SUMMARY:
This is a small pilot intervention tria lfor exercise and air pollution.

DETAILED DESCRIPTION:
This is a pilot randomized, control, clinical trial.

We will recruit 24 adults in Buffalo and randomize them to the physical intervention groups. The intervention group will be provided with physical activity courses.

We will follow up all participants until the end of the study.

We will collect their baseline information via questionnaire, and at the end of the follow-up we will collect the exit questionnaire and biospecimen.

The study aims to demonstrate our ability to recruit eligible participants and provide data of the compliance of participants to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* age 35-55 years old
* plan to stay in Buffalo most of the time in the next three months
* no adverse conditions

Exclusion Criteria:

• those with unstable or life-threatening medical conditions

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-25 (Actual); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
blood pressure | 3 months
  blood pressure will be measured

SECONDARY OUTCOMES:
Self-report questionnaire | 3 months
  This includes how participants feel about the intervention program

CONTACTS AND LOCATIONS:
Overall Officials: Lina Mu, MD,PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States